

## HAROKOPIO UNIVERSITY

## SCHOOL OF HEALTH SCIENCE AND EDUCATION DEPARTMENT OF NUTRITION AND DIETETICS

## **INTERVENTIONTAL STUDY WITH TITLE:**

"Effect of a dietary intervention that includes daily consumption of a novel biscuit enriched with Greek edible mushrooms, rich in β-glucans, on intestinal health-related parameters of healthy older adults: a randomized controlled trial"

## **Analysis**

Data will be analyzed by application of parametric and non-parametric tests depending on fulfillment of normality criteria scrutinization of the data. Statistical analysis will be carried out by using repeated-measures analysis of variance, followed by Tukey's test for multiple comparisons. Age and sex will be used as covariates.